CLINICAL TRIAL: NCT00861523
Title: Comparison Between the Treatment of Thiamine and Promethazine for Improving Vomiting and Nausea in Pregnancy
Brief Title: Does Thiamine Help Vomiting and Nausea in Pregnancy?
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties in recruiting patients
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0101-08-EMC
Record Dates: First submitted 2009-02-18; First posted 2009-03-13 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Hyperemesis Gravidarum
Keywords: nausea; vomiting; pregnancy; thiamine; promethazine; nausea and vomiting in pregnancy
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea; Vomiting | interventions — Thiamine; Promethazine

ARMS (2):
- 1. thiamine (Active Comparator): Pregnant women until 12 week of gestation who refer to the ER because of nausea and vomiting and didn't improve after hydration, will receive thiamine IV
  Interventions: Drug: thiamine & promethazine
- 2. promethazine (Active Comparator): Pregnant women until 12 week of gestation who refer to the ER because of nausea and vomiting and didn't improve after hydration, will receive promethazine IV
  Interventions: Drug: thiamine & promethazine

INTERVENTIONS:
Drug: thiamine & promethazine — thiamine 100 mg IV promethazine 25 mg IV

SUMMARY:
There are different treatments for nausea and vomiting in pregnancy. According to the ACOG recommendations, promethazine is the first line of parenteral treatment after oral treatment had failed. Thiamine is given to prevent wernicke encephalopathy. This research try to find out whether thiamine helps the vomiting and nausea as well, by comparing the response to thiamine and promethazine in women who suffer from nausea and vomiting in pregnancy.

DETAILED DESCRIPTION:
* Research groups: pregnant women eho visit the emergency room for nausea and vomiting in pregnancy, pregnancy age 12 weeks or less
* After basic examinations and hydration, the women will randomized to thiamine or promethazine treatment.
* If no improvement is shown, the patient will be treated with the other drug
* The patients will be interviewed on their current visit and every two weeks until 14th week of gestation
* The interview includes medical history and details about their illness, other treatments, hospitalization etc.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women until 12th week of gestation
* The women visit the ER because of nausea and vomiting
* The women didn't received thiamine yet

Exclusion Criteria:

* Pregnant women over 12th week of gestation
* Women that received thiamine before
* women that allergic to the studied drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
the improvement in nausea and/or vomiting after treatment | 2 months after first visit in ER (until 14 week of pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Yfat Kadan, Principal Investigator — haemek medical center
Locations (1):
- Gynecologic department, Haemek medical center, Afula, Israel